CLINICAL TRIAL: NCT03211416
Title: A Phase Ib/ II Study of Sorafenib and Pembrolizumab in Advanced Hepatocellular Cancer (HCC)
Brief Title: Sorafenib Tosylate and Pembrolizumab in Treating Patients With Advanced or Metastatic Liver Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 35316; NCI-2017-01114 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 35316 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2017-07-05; First posted 2017-07-07 (Actual); Results first posted 2024-05-29 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Advanced Adult Hepatocellular Carcinoma; Child-Pugh Class A; Stage III Hepatocellular Carcinoma; Stage IIIA Hepatocellular Carcinoma; Stage IIIB Hepatocellular Carcinoma; Stage IIIC Hepatocellular Carcinoma; Stage IV Hepatocellular Carcinoma; Stage IVA Hepatocellular Carcinoma; Stage IVB Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — pembrolizumab; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (sorafenib tosylate, pembrolizumab) (Experimental): Patients receive sorafenib tosylate PO BID on days -28 to -1 and 1-21. Patients also receive pembrolizumab IV over 30 minutes on day 1. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: Pembrolizumab; Drug: Sorafenib Tosylate

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475
Drug: Sorafenib Tosylate — Given PO
  Other Names: BAY 43-9006 Tosylate; BAY 54-9085; Nexavar; sorafenib

SUMMARY:
This phase Ib/II trial studies how well sorafenib tosylate and pembrolizumab work in treating patients with liver cancer that has spread to other parts of the body. Sorafenib tosylate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Monoclonal antibodies, such as pembrolizumab, may interfere with the ability of tumor cells to grow and spread. Giving sorafenib tosylate and pembrolizumab may work better in treating patients with liver cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the overall response rate (ORR) related to the combination of sorafenib tosylate (sorafenib) + pembrolizumab in advanced hepatocellular carcinoma patients.

SECONDARY OBJECTIVES:

I. To assess time to tumor progression in patients who received the combination therapy of sorafenib + pembrolizumab compared to historical data on sorafenib only treatment in patients with advanced hepatocellular carcinoma.

TERTIARY OBJECTIVES:

I. To obtain data on changes in immune cell function and in the tumor microenvironment pre- and post-treatment to screen for potential biomarkers that may be able to predict clinical benefit.

- All patients will be followed for survival

OUTLINE:

Patients receive sorafenib tosylate orally (PO) twice daily (BID) on days -28 to -1 and 1-21. Patients also receive pembrolizumab intravenously (IV) over 30 minutes on day 1. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days, every 3 months for up to 1 year, then every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have histologically or radiographically confirmed hepatocellular cancer (HCC) that is advanced or metastatic and if archival tissue is available, have archival tissue submitted for PD-L1, PD-L2 testing
* Participants with measurable disease that has progressed are eligible if prior surgery or locoregional therapy occurred > 28 days prior to enrollment
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0-1 (Karnofsky >= 60%)
* Child-Pugh class-A liver function
* Absolute neutrophil count (ANC) >= 1,500/ mcL
* Hemoglobin >= 8.5 g/dL
* Platelets >= 75,000/ mcL
* Total bilirubin =< 2.0 mg/dL
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 5 X ULN
* Serum Creatinine <= 1.5 upper limit of normal (ULN)or Creatinine clearance > 50 mL/minute if serum creatinine is elevated above 1.5 X ULN
* Have measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria present
* Ability to swallow and retain oral medication
* Participants of child-bearing potential must agree to use adequate contraceptive methods (e.g., hormonal or barrier method of birth control; abstinence) prior to study entry; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Participant must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure
* Participants with past or ongoing hepatitis C virus (HCV) infection will be eligible for the study. The treated participants must have completed their treatment at least 1 month prior to starting study intervention.
* Participants with controlled hepatitis B will be eligible as long as they meet the following criteria:

Antiviral therapy for HBV must be given for at least 12 weeks and HBV viral load must be less than 100 IU/ml prior to first dose of study drug. Participants on active HBV therapy with viral loads under 100 IU/mL should stay on the same therapy throughout study treatment Participants who are anti-HBc , negative for Hepatitis B surface antigen (HBsAg) and negative or positive for anti-HBs, and who have an HBV viral load under 100 IU/mL , do not require HBV anti-viral prophylaxis

Exclusion Criteria:

* One prior line of therapy that may include a PDL1 blocker allowed, no prior sorafenib or PD1 blocker allowed.
* Participants who have had radiotherapy or chemotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Any evidence of bleeding diathesis (patients on therapeutic warfarin or heparin will be excluded)
* Participants with a history of variceal bleed within 6 months prior to enrollment
* Known human immunodeficiency virus (HIV)-positive participants (even if on combination retrovirals, participant will be excluded
* Participants with chronic autoimmune disease
* Participants with known brain metastases should be excluded from this clinical trial
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Has known history of, or any evidence of active, non-infectious pneumonitis
* Pregnant or nursing female participants
* Unwilling or unable to follow protocol requirements
* Any condition which in the Investigator's opinion deems the participant an unsuitable candidate to receive study drug
* Received a live vaccine within 30 days prior to start of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2017-12-07 (Actual); Primary Completion 2023-03-07 (Actual); Study Completion 2025-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kannan Thanikachalam, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (2):
- United States (2):
  - Robert H Lurie Comprehensive Cancer Center, Chicago, Illinois
  - Roswell Park Cancer Institute, Buffalo, New York

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Sorafenib Tosylate, Pembrolizumab)
Started | 37
Completed | 27
Not Completed | 10
Not completed — Adverse Event | 7
Not completed — Lack of Efficacy | 2
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Sorafenib Tosylate, Pembrolizumab)
Number analyzed (Participants) | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.4 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 26
  More than one race | 0
  Unknown or Not Reported | 6
Region of Enrollment [Number; unit: participants]
  United States | 37
Body Mass index [Mean (Standard Deviation); unit: kg/m^2] | 28.5 (5.3)

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate Defined as Partial or Complete Response Per Immune-related Response Evaluation Criteria in Solid Tumors
Description: The response rate will be estimated as the binomial proportion of responders among evaluable patients, and supported by Jeffreys? 95% confidence interval.
Time Frame: Up to 6 months
Population: 10 subjects were not evaluable for response.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Sorafenib Tosylate, Pembrolizumab)
Number analyzed (Participants) | 27
Participants
  Responder (CR+PR) | 8
  non-Responder (SD+PD) | 19
Statistical Analysis 1: Comparison: Treatment (Sorafenib Tosylate, Pembrolizumab); Test type: Superiority; Response Rate = 0.296, 95% CI 2-sided [0.151 to 0.483]

2. Secondary Outcome: Overall Survival
Description: Will be estimated using the Kaplan-Meier method.
Time Frame: From the date of study enrollment to the time of death from any cause, assessed up to 3 year
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Sorafenib Tosylate, Pembrolizumab)
Number analyzed (Participants) | 37
months | 17.1 [6.2 to 37.2]

3. Secondary Outcome: Time to Tumor Progression
Description: Will be estimated using the Kaplan-Meier method, where the median will be estimated with a 95% confidence interval.
Time Frame: From the date of study enrollment to the first observation of progressive disease, assessed up to 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Sorafenib Tosylate, Pembrolizumab)
Number analyzed (Participants) | 37
months | 3.7 [2.5 to 8.7]

4. Other Pre Specified Outcome: Change in Functional Activity of Effector T Cells
Description: The effect of treatment will be quantified as the post/pre-treatment mean ratio of the expression measurements, assessed using a two-sided one sample t-test.
Time Frame: Up to 3 years
Population: Only 20 subjects had paired pre-treatment and post-treatment flow data available.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Treatment (Sorafenib Tosylate, Pembrolizumab)
Number analyzed (Participants) | 20
ratio | 1.17 (0.84)
Statistical Analysis 1: Comparison: Treatment (Sorafenib Tosylate, Pembrolizumab); The null hypothesis is that the mean ratio of T effect cells (post / pre) is equal to 1 (no change); Test type: Superiority; p = 0.40, Two-sided, one-sample t-test — Significance level of 0.05

5. Other Pre Specified Outcome: Change in Levels of Immunosuppressive Cells
Description: as for outcome 4
Time Frame: Up to 3 years
Population: Data was not captured.
Arm/Group | Treatment (Sorafenib Tosylate, Pembrolizumab)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were followed for up to 30 days post-treatment initiation, which was a median of 140 days (range = 41 to 1,162 days). All cause mortality was monitored for up to 3 years following treatment initiation.
Arm/Group | Treatment (Sorafenib Tosylate, Pembrolizumab)
All-Cause Mortality (participants affected / at risk) | 24/37
Serious Adverse Events (participants affected / at risk) | 20/37
Other Adverse Events (participants affected / at risk) | 36/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Sorafenib Tosylate, Pembrolizumab) (N=37)
Aortic valve disease (Cardiac disorders) | 1 (1)
Heart failure (Cardiac disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Duodenal hemorrhage (Gastrointestinal disorders) | 1 (1)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1)
Death NOS (General disorders) | 3 (3)
Fever (General disorders) | 1 (1)
Multi-organ failure (General disorders) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 2 (2)
Immune system disorders - Other (Immune system disorders) | 4 (4)
Appendicitis perforated (Infections and infestations) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 1 (1)
Infections and infestations - Other (Infections and infestations) | 2 (2)
Sepsis (Infections and infestations) | 3 (3)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Sorafenib Tosylate, Pembrolizumab) (N=37)
Anemia (Blood and lymphatic system disorders) | 3 (3)
Hypothyroidism (Endocrine disorders) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 8 (8)
Constipation (Gastrointestinal disorders) | 5 (5)
Diarrhea (Gastrointestinal disorders) | 23 (23)
Mucositis oral (Gastrointestinal disorders) | 4 (4)
Nausea (Gastrointestinal disorders) | 8 (8)
Vomiting (Gastrointestinal disorders) | 3 (3)
Chills (General disorders) | 6 (6)
Edema limbs (General disorders) | 3 (3)
Fatigue (General disorders) | 21 (21)
Fever (General disorders) | 4 (4)
Alanine aminotransferase increased (Investigations) | 4 (4)
Aspartate aminotransferase increased (Investigations) | 7 (7)
Blood bilirubin increased (Investigations) | 9 (9)
Lymphocyte count decreased (Investigations) | 3 (3)
Weight loss (Investigations) | 13 (13)
Anorexia (Metabolism and nutrition disorders) | 20 (20)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 9 (9)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Dizziness (Nervous system disorders) | 4 (4)
Dysgeusia (Nervous system disorders) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (4)
Dry skin (Skin and subcutaneous tissue disorders) | 6 (6)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 16 (16)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 11 (11)
Hypertension (Vascular disorders) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-30): https://cdn.clinicaltrials.gov/large-docs/16/NCT03211416/Prot_SAP_000.pdf